CLINICAL TRIAL: NCT01228786
Title: Transcriptional and Translational Regulation of Vitamin D Receptor (VDR) and Calcium Sensing Receptor (CaSR) in Patients With Sporadic Primary Hyperparathyroidism
Brief Title: Regulation of Vitamin D Receptor (VDR),Calcium Sensing Receptor (CaSR), Cyclin D1,Ki67 and Proliferating Cell Nuclear Antigen (PCNA) in Primary Hyperparathyroidism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sanjay K. Bhadada, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Other Study IDs: BHADADA-PGI; BHADADA-SK (Other: ICMR, India)
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Primary Hyperparathyroidism (PHPT)
Keywords: VDR, CaSR, PTH, Cyclin D1, Ki67, PCNA
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Parathyroid Adenoma and normal parathyroid gland
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: ~ 20 sporadic PHPT patients
- Group B: ~10 normocalcemic euthyroid patients (control tissue)

SUMMARY:
The present study is designed to examine the expression of VDR, CaSR, PTH, Cyclin D1, Ki67 and PCNA and to find out its relationship with clinical parameters in parathyroid adenomas. Examination of the contribution of genes expression can elucidate the critical link between proliferation and functional abnormalities in parathyroid adenomas. Alternative to DNA and RNA, protein expression can provide a better understanding of this disease.

DETAILED DESCRIPTION:
Introduction:

Primary hyperparathyroidism (PHPT) is the third most frequent endocrine disorder, after diabetes mellitus and thyroid disorders, that predominantly affects postmenopausal women, with an incidence of 1 -5 in 1000 people. It can occur at any age though young people are rarely affected. PHPT is characterized by hypersecretion of parathyroid hormone (PTH) and resultant hypercalcemia. Most cases of PHPT (>85%) result from a solitary adenoma in one of the parathyroid glands. Multi-gland hyperplasia is found in about 10-15% of the patients while carcinoma occurs rarely (1-2%).

The parathyroid glands regulate calcium homeostasis. The major target organs for parathyroid hormone (PTH) are bone and the kidneys. PTH increases bone resorption to mobilize calcium into the circulation. In the kidney, PTH enhances calcium reabsorption and increases phosphate excretion. PTH also stimulates renal production of 1α,25-dihydroxyvitamin D [1,25(OH)2D], which in turn enhances intestinal absorption of calcium. Thus, the physiological effects of PTH are to increase the concentration of calcium in the circulation. Negative feedback from calcium and 1,25(OH)2D modulate parathyroid function. These effects are mediated via the calcium-sensing receptor (CaSR) expressed on the parathyroid cell surface. Similarly, 1,25(OH)2D, acts through vitamin D receptor (VDR) and suppresses PTH synthesis and secretion . Thus, PTH secretion is tightly coupled to the parathyroid cell's ambient calcium level.

Increased parathyroid cell proliferation and decreased calcium-mediated control of the PTH secretion are characteristic findings in all types of hyperparathyroidism (1-4). Calcium via its receptor, the CaSR and the 1,25(OH)2D-VDR complex are the most important regulators, in this respect. Decreased actions of these regulators would stimulate the parathyroid cells to proliferate. Molecular analyses have revealed the presence of tumor-specific DNA rearrangements in a subset of adenomas. In such rearrangements, the 5' PTH gene regulatory region combines upstream of the Cyclin D1 gene, which results in over expression of cyclins that could induce proliferation by increasing mitotic rate. In fact Cyclin D1 over expression was first demonstrated in a patient with parathyroid adenoma (5).

Impaired CaSR gene expression is found in parathyroid lesions of both primary and secondary hyperparathyroidism (6-11). No mutations could be found in CaSR gene in parathyroid neoplasias (11,12). Similar present findings shows reduced VDR gene expression (8,13-15) and concur with studies on the apparent lack of VDR gene mutations in hyperparathyroidism (16-18). Differential expression of VDR and CaSR gene has been reported in a few parathyroid adenomas, but exact mechanism is not known. These observations raise the possibility that altered expression of these genes could be related to the pathogenesis of parathyroid adenomas.

OBJECTIVES: To achieve the above aim, the following objectives would be under taken.

1. Comparison of expression of VDR and CaSR genes in parathyroid adenomas with normal parathyroid tissue obtained during surgery from non-hyperparathyroid patients by Real Time-PCR.
2. To confirm expression of VDR, CaSR,PTH cyclin D1, Ki67 and PCNA in parathyroid cells by immunohistochemistry.
3. Comparison of protein expression profile of parathyroid adenomas with normal parathyroid tissue by proteomic analysis.

MATERIALS AND METHODS:

Subjects:

All the PHPT patients attending outdoor patient clinic of Endocrinology and General Surgery department of Nehru Hospital, PGIMER, Chandigarh will be included for this study with following inclusion and exclusion criteria.

Inclusion Criteria: Patients with surgically verified sporadic PHPT and controls will be included as follows; Group A: ~ 20 sporadic PHPT patients Group B: ~10 normocalcemic euthyroid patients operated for thyroid disorders will provide normal parathyroid tissue to serve as control tissue.

Exclusion Criteria: Patients with hyperplasia, renal failure and multiple endocrine neoplasia will be excluded.

Sample collection: Parathyroid tissue samples will be collected immediately after surgery, snap frozen and stored at -80oC until use.

Assay Methods: Preoperative levels of total serum calcium (reference range, 8.6-10.2 mg/dL) will be determined by auto-analyzer (Modular P: Roche Diagnostics, Germany). The serum Calcium level will be corrected with the serum albumin level. The serum intact PTH (reference range, 12-55 ng/L)and 25-hydroxyvitamin D (11.1-42.9 ng/ml) will be measured using immunochemiluminiscence (ELECSYS-2010: Roche Diagnostics, Germany).

1. Gene expression study for VDR and CaSR-

   1. RNA extraction:

      Total RNA will be extracted from the cryopreserved normal and adenomatous parathyroid tissue samples by using the TRIZOL reagent (Life Technologies, Inc.), according to the vendor's instructions. The samples will be pretreated with DNase and stored at -80oC until use. The cDNA will be generated from the 3-4 mg of RNA by reverse transcriptase with random hexamers as primers.
   2. Real-Time Polymerase Chain Reaction:

   The mRNA levels of VDR and CaSR will be estimated by Real-PCR (Stratagene Robocycler Gradient 40 system) using specific primer sequences and PCR conditions. The PCR products will be separated by electrophoresis on 6% agarose gel; the products will be then stained with ethidium bromide and located by fluorescence using UV light. Bio Max 1D TM 1.5.1 (Kodak, Rochester, NY) would be used to evaluate the band intensities of the PCR bands.
2. Expression study of VDR, CaSR,PTH, Cyclin D1, Ki67 and PCNA protein-

   Immunohistochemistry: Monoclonal antibodies will be used for immunostaining of VDR, CaSR, PTH, Cyclin D1, Ki67 and PCNA proteins on paraffin sections (Source- Pharmingen, USA). Secondary antibody, goat anti-mouse horse radish peroxidase conjugated (BD Biosciences, Pharmingen, USA), specific for primary antibodies will be used in each test. Indirect immunoperoxidase method will be used for the staining of paraffin sections. In this assay, the unconjugated primary antibody binds to the antigen in the specimen. To localize this attachment, a peroxidase conjugated specific secondary antibody is used which binds to the primary antibody. A substrate is than added to localize the reaction.

   The slides will be then examined under the light microscope. Staining will be graded as negative (0), mild (+), moderate (++) and marked (+++) depending on intensity of immunoreactivity.
3. Comparison of protein expression profile-

   1. Extraction of Proteins 100mg of tissue will be homogenized with 0.5 ml of cold (4°C) lysis buffer. Protein will be estimated by Bicin chronic Acid (BCA) method and store the remaining at -80°C.
   2. First Dimension (IEF) and Second Dimension (SDS-PAGE) separation The concentrated sample will be solubilized in rehydration buffer. A total 125 - 200 µl will be loaded onto 7 cm IPG strip (Amersham). IEF run will be according to manufacturer's protocol.

      For second dimension the IPG strips will be equilibrated for 15 min with 6 ml equilibration buffer. Each IPG strip will be loaded onto 12% polyacrylamide gel and electrophoresed (100 or 200 V for ~6 h). After electrophoresis, proteins will be fixed and are visualized using Coomassie and Silver stains.
   3. Image Analysis, In-gel trypsin digestion and MALDI mass spectrometry analysis Stained gels will be scanned with GS-800 densitometer (Bio-Rad) using PDQuest software (Bio-Rad) and the proteins of interest will be analyzed by the MALDI-TOFMS (Voyager DE-PRO, Applied Biosystems) at Institute of microbial technology (IMTech).

Proteins will be identified by peptide mass fingerprinting using Mascot web based Search engine with the help of peptide mass spectra.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgically verified sporadic PHPT

Exclusion Criteria:

* Patients with hyperplasia, renal failure and multiple endocrine neoplasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Primery Hyperparathyroidism (PHPT)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sanjay K. Bhadada, DM, Principal Investigator — Indian Counsil of Medical Research
Locations (1):
- PGIMER, Chandigarh, Uttarakhand, India